CLINICAL TRIAL: NCT00619268
Title: Open Label, Randomized, Multicenter Phase II Study of a Combination of Torisel® (Temsirolimus) and Avastin® (Bevacizumab) Versus Sutent® (Sunitinib) and Versus a Combination of Avastin® (Bevacizumab) and Roféron® (Interferon Alpha-2a) in First-line Treatment of Patients With Metastatic Renal Cell Carcinoma.
Brief Title: Combination of Temsirolimus and Bevacizumab in Patient With Metastatic Renal Cell Carcinoma
Acronym: TORAVA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TORAVA; ET2007-035
Record Dates: First submitted 2008-02-08; First posted 2008-02-20 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Metastatic Renal Cell Carcinoma
Keywords: Temsirolimus; Bevacizumab; Metastatic renal cell carcinoma; Non-progression
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — temsirolimus; Bevacizumab; Sunitinib; Interferon alpha-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A (Experimental)
  Interventions: Drug: Temsirolimus; Drug: Bevacizumab
- B (Active Comparator)
  Interventions: Drug: Sunitinib
- C (Active Comparator)
  Interventions: Drug: Bevacizumab; Drug: Interferon alpha-2a

INTERVENTIONS:
Drug: Temsirolimus — 25 mg once per week administered intravenously
  Other Names: Torisel®
  Arms: A
Drug: Bevacizumab — 10 mg/kg * 1 time /2 weeks administered intravenously
  Other Names: Avastin®
  Arms: A; C
Drug: Sunitinib — 50 mg administered orally once daily in 6 weeks cycles :4 weeks of treatment followed by 2 weeks off
  Other Names: Sutent®
  Arms: B
Drug: Interferon alpha-2a — Administered subcutaneously as 9 MU three times per week
  Other Names: Roféron®
  Arms: C

SUMMARY:
The TORAVA trial is designed to evaluate the progression-free rate at 48 weeks of a combination of Torisel® and Avastin® given at first-line treatment in patients with metastatic renal cancer.

Eligible patients will be randomly assigned, in a 2:1:1 ratio, to either Avastin® + Torisel®, or Sutent® or IFN+Avastin®.

DETAILED DESCRIPTION:
This is a phase II, open label, randomized, parallel group, multicenter study evaluating first-line treatment of patients with metastatic renal cancer using a combination of Torisel® administered intravenously as 25 mg every week and Avastin® administered intravenously as 10 mg/kg every 2 weeks.

Two standard arms with either Sutent® (given orally as 50 mg once daily during 4 weeks, followed by 2 weeks off) or a combination of Avastin® (administered intravenously as 10 mg/kg every 2 weeks) and Interferon (IFN, administered subcutaneously as 9 MU three times a week) will be used to validate the results obtained in the experimental arm (randomization eliminates selection biases), and to assess Sutent® efficacy rate on a more representative population than in Motzer's trial (Motzer NEJM 2007).

The study is not designed to provide head-to-head comparisons between the experimental arm (Avastin® + Torisel®) and the two standard arms (Sutent® and IFN + Avastin®). Randomization will be used as a tool for allocating patients evenly into the 3 treatment arms to ensure proper balance of prognostic factors. If the progression-free rates observed in randomly assigned control patients are inconsistent with historical data, it may be a warning that the results observed for the experimental arm should be viewed with caution. Patients will be randomly assigned to either option in a 2:1:1 ratio (half less patients in the standard arms used only as historical comparators), and stratified according to inclusion center and performance status (ECOG PS 0 vs. 1 vs. 2).

In the absence of severe toxicity, treatment will be continued until documented progression of the disease (RECIST criteria). Toxicity will be evaluated throughout the treatment period and until disappearance or stabilization of the side effect(s). In case of progression, each investigator makes his/her own treatment decisions, provided that all anti-cancer treatments given to the patients within the frame of the study are reported, as well as their results.

Response rates will be assessed between weeks 11-12, 23-24, 35-36, 47-48 in the first year (corresponding to 2 cycles of Sutent®) and every 3 months afterwards until treatment stop, or until patient death or end of clinical data collection.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients>= 18 years of age;
* Patients with histological or cytological evidence of metastatic renal cell carcinoma mostly of all type,except for papillary;
* No prior systemic treatment (chemotherapy, immunotherapy, anti-angiogenic drugs, or treatment under evaluation) for metastatic renal cancer;
* No brain metastases revealed by MRI or CT-scan within 28 days prior to randomization. Patients with a history of brain metastases treated by surgery +/- radiation therapy can be included if they have normal brain MRI;
* E.C.O.G performance status =<2;
* At least one measurable lesion using the RECIST criteria;
* Blood tests and renal and liver functions in the normal range with, in the 7 days prior to study entry, blood or serum values as follows:

Hemoglobin > 8g/dl; Neutrophil count > 1500*10exp9/L; Platelets > 100*10exp9/L; Serum creatinine < 200µmol/L; Total Bilirubin < 1.5 times upper limit of normal; ALT and AST < 2.5 times upper limit of normal or < 5 ULN for patients with liver metastases, PT or INR < 1.5 times upper limit of normal in the absence of anticoagulant therapy;

* Absence of proteinuria confirmed by urinary dipstick test
* Fertile women must use effective means of contraception
* Mandatory affiliation with a healthy security insurance
* Signed written informed consent.

Exclusion Criteria:

* Patient with pure papillary renal cell carcinoma
* Prior systemic treatment for metastatic renal cancer
* History of other malignancies, other than curatively treated in-situ carcinoma of the cervix or basal cell carcinoma of the skin, or any other curatively treated cancer with no sign of recurrence within 5 years prior to randomization
* Evidence of brain metastasis by computerized tomographic scan or MRI in the 28 days prior to randomization. Patients with history of brain metastases treated by exclusive brain therapy are not allowed to participate, even if brain MRI is normal
* Significant cardiovascular disease or uncontrolled hypertension while receiving appropriate medication (>= 160 mm Hg systolic and/or >= 90 mm Hg diastolic)
* Hepatic affection like chronic advanced hepatitis, liver cirrhosis or chronic hepatitis recently treated or in process of treatment by immunosuppressive agents, hepatitis auto-immune or history of auto-immune disease
* Major surgical procedure, open biopsy, or serious non healing wound within 28 days prior to randomization
* Uncontrolled hypercalcemia while receiving appropriate treatment
* Uncontrolled hypercholesterolemia or hypertriglyceridemia
* Patient under anti-vitamin K therapy
* Patient under strong CYP3A4 inhibitors
* Patient with severe neuropsychiatric disorder (or comitial crises)
* Patient included in another clinical trial, except for supportive care trials
* Pregnant or lactating women (mandatory negative serum or urinary pregnancy test at study entry for all women of childbearing potential)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2008-02; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
progression-free rate | at 48 weeks post-treatment

SECONDARY OUTCOMES:
Objective response rate:efficacity | Every 12 weeks during 48 weeks
Duration of response
Toxicity | at week 2, week 5-6 and after every 5-6 weeks during 48 weeks
Quality of life | at inclusion, month 6 and at 1 year
progression-free survival and overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie NEGRIER, MD, PhD, Principal Investigator — Centre Leon Berard; Bernard ESCUDIER, MD, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (29):
- France (29):
  - Centre Paul Papin, Angers
  - Centre Hospitalier Universitaire de Besançon, Besançon
  - Centre Hospitalier Universitaire de Bordeaux - Hôpital St André, Bordeaux
  - Institut Bergonié, Bordeaux
  - Centre François Baclesse, Caen
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Georges François Leclerc, Dijon
  - Centre Hospitalier de Versailles, Le Chesnay
  - Centre Hospitalier Universitaire de Lille - Hôpital Claude Huriez, Lille
  - Centre Oscar Lambret, Lille
  - Centre Hospitalier Universitaire DUPUTRYEN, Limoges
  - Centre Léon Bérard, Lyon
  - Centre Hospitalier Universiariare Lyon, Hôpital Lyon Sud, Lyon
  - Institut Paoli Calmette, Marseille
  - Centre Val d'Aurelle, Montpellier
  - Clinique Valdegour-Centre médical Oncogard, Nîmes
  - Fondation Hôpital Saint Joseph, Paris
  - Hopital du Val de Grâce, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - Centre Hospilier Universitaire de Poitiers, Poitiers
  - Institut Jean Godinot, Reims
  - Centre Eugène Marquis, Rennes
  - Centre René Gauducheau, Saint-Herblain
  - Institut de Cancérologie de la Loire, Saint-Priest-en-Jarez
  - Centre Hospitalier Starsbourg, Strasbourg
  - Hôpital FOCH, Suresnes
  - Institut Claudius Regaud, Toulouse
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif

REFERENCES:
- [Background] Escudier B, Eisen T, Stadler WM, Szczylik C, Oudard S, Siebels M, Negrier S, Chevreau C, Solska E, Desai AA, Rolland F, Demkow T, Hutson TE, Gore M, Freeman S, Schwartz B, Shan M, Simantov R, Bukowski RM; TARGET Study Group. Sorafenib in advanced clear-cell renal-cell carcinoma. N Engl J Med. 2007 Jan 11;356(2):125-34. doi: 10.1056/NEJMoa060655. PMID 17215530
- [Background] Motzer RJ, Hutson TE, Tomczak P, Michaelson MD, Bukowski RM, Rixe O, Oudard S, Negrier S, Szczylik C, Kim ST, Chen I, Bycott PW, Baum CM, Figlin RA. Sunitinib versus interferon alfa in metastatic renal-cell carcinoma. N Engl J Med. 2007 Jan 11;356(2):115-24. doi: 10.1056/NEJMoa065044. PMID 17215529
- [Background] Hudes G, Carducci M, Tomczak P, Dutcher J, Figlin R, Kapoor A, Staroslawska E, Sosman J, McDermott D, Bodrogi I, Kovacevic Z, Lesovoy V, Schmidt-Wolf IG, Barbarash O, Gokmen E, O'Toole T, Lustgarten S, Moore L, Motzer RJ; Global ARCC Trial. Temsirolimus, interferon alfa, or both for advanced renal-cell carcinoma. N Engl J Med. 2007 May 31;356(22):2271-81. doi: 10.1056/NEJMoa066838. PMID 17538086
- [Result] Negrier S, Gravis G, Perol D, Chevreau C, Delva R, Bay JO, Blanc E, Ferlay C, Geoffrois L, Rolland F, Legouffe E, Sevin E, Laguerre B, Escudier B. Temsirolimus and bevacizumab, or sunitinib, or interferon alfa and bevacizumab for patients with advanced renal cell carcinoma (TORAVA): a randomised phase 2 trial. Lancet Oncol. 2011 Jul;12(7):673-80. doi: 10.1016/S1470-2045(11)70124-3. Epub 2011 Jun 12. PMID 21664867
- [Derived] Aldin A, Besiroglu B, Adams A, Monsef I, Piechotta V, Tomlinson E, Hornbach C, Dressen N, Goldkuhle M, Maisch P, Dahm P, Heidenreich A, Skoetz N. First-line therapy for adults with advanced renal cell carcinoma: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 May 4;5(5):CD013798. doi: 10.1002/14651858.CD013798.pub2. PMID 37146227
- [Derived] Polena H, Creuzet J, Dufies M, Sidibe A, Khalil-Mgharbel A, Salomon A, Deroux A, Quesada JL, Roelants C, Filhol O, Cochet C, Blanc E, Ferlay-Segura C, Borchiellini D, Ferrero JM, Escudier B, Negrier S, Pages G, Vilgrain I. The tyrosine-kinase inhibitor sunitinib targets vascular endothelial (VE)-cadherin: a marker of response to antitumoural treatment in metastatic renal cell carcinoma. Br J Cancer. 2018 May;118(9):1179-1188. doi: 10.1038/s41416-018-0054-5. Epub 2018 Mar 22. PMID 29563634